CLINICAL TRIAL: NCT06939894
Title: The Effects of Drama Activities on Nursing Students' Attitudes Towards Pain Assessment: A Randomised Controlled Trial
Brief Title: The Effects of Drama Activities on Nursing Students' Attitudes Towards Pain Assessment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Gulden Basit, Assoc. Prof., Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NEU-GB-OB-1
Record Dates: First submitted 2025-04-11; First posted 2025-04-23 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Pain Assessment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): no intervention, usual curriculum.
- Drama (Experimental): will take drama activities
  Interventions: Behavioral: Drama activities

INTERVENTIONS:
Behavioral: Drama activities — iintervention group will paticipate drrama activities aabout pain assessment of a patient.
  Arms: Drama

SUMMARY:
Title:

The Effect of Drama-Based Education on Nursing Students' Attitudes Toward Pain Assessment: A Randomized Controlled Trial

Abstract:

This randomized controlled trial aims to investigate the effect of drama-based education on nursing students' attitudes toward pain assessment. The study will be conducted during the 2025-2026 academic year at Necmettin Erbakan University, Faculty of Nursing. A total of 52 second-year students who meet the inclusion criteria will be randomly assigned to intervention and control groups.

The intervention group will attend a one-day drama workshop involving role-play, improvisation, and reflection activities focused on pain assessment. The control group will not receive any intervention. Attitudes will be measured using a validated scale at three points: before the intervention, one month after, and six months after.

Data will be analyzed using SPSS with a significance level of p < 0.05. It is anticipated that the intervention group will show improved attitudes compared to the control group.

This study may provide evidence for integrating drama-based methods into nursing education to enhance students' sensitivity and competence in pain assessment.

Keywords:

Nursing education, pain assessment, drama, student attitudes,

DETAILED DESCRIPTION:
This study is designed as a randomized controlled trial using a pretest-posttest design to examine the effect of drama-based education on nursing students' attitudes toward pain assessment. The research will be conducted during the 2025-2026 academic year at the Faculty of Nursing, Necmettin Erbakan University (NEU), which offers education in nine nursing departments. The study population consists of second-year nursing students (n=160). The sample will include students whose native language is Turkish, who have not received any formal education in pain management, and who volunteer to participate. Sample size was calculated using G*Power 3.1.9.2, based on Cohen's conventional effect size (d=0.80, power=0.80, two sided), resulting in a total of 52 students (26 in each group), allowing for potential attrition.

Participants will be randomly assigned to intervention and control groups via random.org by an independent statistician. Data will be collected face-to-face using a Descriptive Information Form and the Attitudes of Nursing Students Toward Pain Assessment Scale. The intervention group will participate in a one-day drama-based workshop designed by a certified drama leader, focusing on pain assessment. The attitude scale will be administered before the intervention, one month later (November 2025), and approximately six months later (at 2025-2026 academic year). The control group will complete the same data collection tools at equivalent time points without receiving any intervention.

Drama activities will follow the preparation, enactment, and reflection phases, utilizing techniques such as role-play, improvisation, and pantomime. The dependent variable is the mean attitude score toward pain assessment; the independent variable is the drama activity, while control variables include age, gender, knowledge of pain assessment methods and tools, prior education in pain management, and clinical experience with patients in pain. Data will be analyzed using SPSS software, applying descriptive statistics and appropriate parametric or non-parametric tests based on normality. Significance will be set at p<0.05.

Ethical approval will be obtained from the NEU Scientific Research Ethics Committee and the Faculty of Nursing. Written and verbal informed consent will be collected from all participants. Permission to use the attitude scale has been granted by the original authors. After data collection, the drama intervention will also be offered to the control group to ensure ethical balance.

Keywords: Nursing education, pain assessment, drama-based intervention, student attitudes

ELIGIBILITY:
Inclusion Criteria: The study group will consist of second-year students

* the study sample will consist of students whose native language is Turkish,
* who have not taken a course on pain management,
* and who volunteer to participate in the study.

Exclusion Criteria:

* students who wish to withdraw from research

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2026-04-23 (Estimated); Study Completion 2026-04-23 (Estimated)

PRIMARY OUTCOMES:
pain assessment attitudes of students | Day 0, month 1., and month 6.
  Students will be randomly assigned to the intervention and control groups. Students in the intervention group will fill out the introductory characteristics form and the nursing students' attitudes towards pain assessment scale after being assigned to the group and will then participate in drama activities prepared for pain assessment for one day. The students' attitudes towards pain assessment scale will be filled out again by the students one month after the intervention (November 2025) and approximately six months later (at 2025-2026 academic year). Students in the control group will fill out the introductory characteristics form and scale on the same dates as the experimental group without any intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Gülden Basit, Study Chair — Necmettin Erbakan University
Locations (2):
- Turkey (Türkiye) (2):
  - Necmettin Erbakan University, Meram, Konya
  - Necmettin Erbakan University, Meram